CLINICAL TRIAL: NCT04473248
Title: Evaluation of Clinical Sample Collection Project: Spartan COVID-19
Brief Title: Spartan COVID-19 System: Evaluation of Clinical Sample Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spartan Bioscience Inc. (Industry)
Collaborators: Humber River Hospital (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: VNV-00552
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Each Patient enrolle dint he study will experience the same modes of sample collection and sample analysis.
Who Masked: Participant
Masking Description: The results of the Spartan COVID-19 System tests will not be shared with the participant or the lab, but the lab results will be shared with Spartan once analysis of the Spartan System samples is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Method 1- Nasopharyngeal Swab in transfer liquid (Experimental): A nasopharyngeal swab will inoculate a proprietary solution which will be transferred to the Spartan COVID-19 System for analysis
  Interventions: Device: Spartan COVID-19 System
- Method 2- Dipping of specialized swab in VTM (Experimental): A nasopharyngeal swab will inoculate VTM solution. A modified traditional Spartan Swab will be dipped into the inoculated VTM solution and then transferred to the Spartan COVID-19 System for analysis.
  Interventions: Device: Spartan COVID-19 System
- Method 3: Direct input of VTM (Experimental): Using the VTM from Method 2, pipette 10uL of VTM, inoculated with sample, into the Spartan COVID-19 System for analysis.
  Interventions: Device: Spartan COVID-19 System
- Method 4: Collection of nasal sample. (Experimental): Using a modified tip of the Spartan swab, a nasal sample will be taken from the patient and directly placed into the Spartan COVID-19 System for analysis.
  Interventions: Device: Spartan COVID-19 System

INTERVENTIONS:
Device: Spartan COVID-19 System — PCR analysis of patient samples using the Spartan COVID-19 System

SUMMARY:
This study will evaluate the efficacy of various sample collection methods for use with the Spartan COVID-19 System. It will compare the results from the Spartan COVID-19 System with results that are obtained using a predicate lab-based COVID-19 test that uses a nasopharyngeal swab sample. The goal is to determine which sample collection methods are most effective in capturing SARS-CoV-2 virus.

DETAILED DESCRIPTION:
Once the subject is recruited,two nasopharyngeal swabs using the standard method will be taken from the patient. Additionally, two nasal swab samples will be taken using the Spartan COVID-19 swabs with an adjusted tip. All samples will be analyzed using the Spartan COVID-19 System.

The lab-based predicate test will be taken at the same time, with results reported back to Spartan to be compared with results obtained from the Spartan COVID-19 System.

ELIGIBILITY:
Inclusion Criteria:

* must have tested positive for COVID-19 via the existing nucleic acid testing method.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Asses the % agreement between predicate results and Spartan COVID-19 results. | Through study completion; anticipated to be less than 6 months.
  The purpose of this study is to evaluate which method has the best % agreement between the lab-based predicate results and Spartan COVID-19 System results.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Linseman, MSc, Study Director — Spartan Bioscience Inc.
Locations (2):
- Canada (2):
  - Humber River Hospital, North York, Ontario
  - The Univeristy of Ottawa Heart Institute, Ottawa, Ontario